CLINICAL TRIAL: NCT05746650
Title: Regulation of Protein Turnover in Connective Tissue From Muscle and Tendon Following Muscle Tissue Injury
Brief Title: Improving Tissue Repair After Injury in the Muscle-tendon Interface Muscle Tissue Injury
Acronym: GH-MTJ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Grith Højfeldt, Principal Investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BBH158
Record Dates: First submitted 2023-01-24; First posted 2023-02-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Muscle Injury
MeSH Terms: interventions — Electric Stimulation; Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1) Electrical stimulation + growth hormone (Experimental): One bout of electrical stimulation with 200 eccentric contractions. This is followed by daily injections with somatropin (33.3 ug/kg in the first week, 50 ug/kg in the second week) for two weeks.
  Interventions: Procedure: Electrical stimulation; Drug: Growth hormone (somatropin)
- 2) Electrical stimulation (Experimental): One bout of electrical stimulation with 200 eccentric contractions
  Interventions: Procedure: Electrical stimulation
- 3) Growth hormone (Active Comparator): Daily injections with somatropin (33.3 ug/kg in the first week, 50 ug/kg in the second week) for two weeks.
  Interventions: Drug: Growth hormone (somatropin)
- 4) Control (Placebo Comparator): No intervention
  Interventions: Other: Control (No electrical stimulation, nor growth hormone)

INTERVENTIONS:
Procedure: Electrical stimulation — Experimentally induced muscly injury via. neuromuscular electrical stimulation of the hamstring muscles
  Arms: 1) Electrical stimulation + growth hormone; 2) Electrical stimulation
Drug: Growth hormone (somatropin) — Daily injection of growth hormone
  Arms: 1) Electrical stimulation + growth hormone; 3) Growth hormone
Other: Control (No electrical stimulation, nor growth hormone) — No electrical stimulation, nor growth hormone
  Arms: 4) Control

SUMMARY:
The study is a 2-week human study where 40 patients who are scheduled to undergo reconstructive knee surgery are randomized to administration of GH or placebo following or without neuromuscular electrical stimulation of hamstring muscles.The overall aim is to determine, the role of muscle connective tissue protein synthesis in muscle injury and repair.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women scheduled to undergo reconstructive knee surgery
* BMI 18-35

Exclusion Criteria:

* Former or current use of growth hormone or anabolic steroids
* Use of corticosteroids in the past 3 months
* Use of any medication known to affect muscle or tendon turnover
* Former participation in a study using deuterated water
* Chronic diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in muscle and myotendinous junction protein synthesis in regenerating vs. control muscle | 2 years
  Fractional synthesis rates based on D2O (deuterated water) intake and deuterium labelled alanine in tissue

SECONDARY OUTCOMES:
Difference in muscle protein synthesis in regenerating muscle, myotendinous junction tissue with or without growth hormone | 2 years
  Fractional synthesis rates based on D2O (deuterated water) intake and deuterium labelled alanine in tissue
Single protein synthesis in regenerating vs. control muscle and myotendinous junction tissue | 2 years
  Dynamic proteome profiling fractional synthesis rates based on D2O (deuterated water) intake and deuterium labelled alanine in single proteins
Single protein synthesis in regenerating muscle and myotendinous junction tissue with or without growth hormone | 2 years
  Dynamic proteome profiling fractional synthesis rates based on D2O (deuterated water) intake and deuterium labelled alanine in single proteins
Tendon tissue synthesis from injured muscle vs. control muscle | 2 years
  FSR based on D2O intake and D-alanine label in tissue
Difference in muscle protein synthesis in regenerating muscle, myotendinous junction, and tendon tissue with or without growth hormone | 2 years
  Fractional synthesis rates based on D2O (deuterated water) intake and deuterium labelled alanine in tissue
Difference in muscle protein synthesis in regenerating vs. control muscle, myotendinous junction, and tendon tissue | 2 years
  Fractional synthesis rates based on D2O (deuterated water) intake and deuterium labelled alanine in tissue
Number of satellite cells, fibroblasts and immune cells in renereting vs. control tissue, with and without growth hormone | 2 years
  Histochemical staining of muscle cross sections
Mechanical properties of tissue with and without growth hormone | 2 years
  Ex vivo mechanical stress test

CONTACTS AND LOCATIONS:
Overall Officials: Grith Højfeldt, PhD, Principal Investigator — Institute of Sports Medicine, Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided